CLINICAL TRIAL: NCT04140370
Title: Frailty Prevalence in Surgical European Patients. European Prospective Cohort Stufy of the Prevalence of Frailty in Surgical Patients.
Acronym: FRAGILE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Spanish Multimodal Rehabilitation Group (Unknown); Spanish Sociey of Anesthesiology (Unknown)
Responsible Party: Principal Investigator, Carlos Ferrando Ortolá, Head of Surgical Intensive Care Unit, Hospital Clinic of Barcelona
Other Study IDs: FRAGILE
Record Dates: First submitted 2019-10-18; First posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: There is no intervention — There is no intervention

SUMMARY:
European prospective one day cohort study. Analysis of the prevalence of frailty and predefined 30-day postoperative complications in adult patients undergoing emergency or elective surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who will undergo emergency or elective surgery with an intended hospital stay of more than 24 hours and any type of anesthesia.

Exclusion Criteria:

* Outpatient (ie. day case) surgery, obstetric analgesia or anesthesia, organ transplant surgery, cardiac surgery, neurosurgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo emergency or elective surgery with an intended hospital stay of more than 24 hours and any type of anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 6500 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2020-08-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with frailty identified in the preoperative assessment in both elective and emergency surgery, as well as frailty's severity. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: César Aldecoa, MD, Principal Investigator — Hospital Río Ortega

IPD SHARING:
Plan to Share IPD: No